CLINICAL TRIAL: NCT02786771
Title: Exploring the Effects of Muse and Spire on Stress Management
Acronym: Stressless
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joseph C. Kvedar, Dermatologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016P000508
Record Dates: First submitted 2016-05-23; First posted 2016-06-01 (Estimated); Results first posted 2018-05-16 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Stress
Keywords: Stress Management; Mindfulness; Meditation; Stress Resilience

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spire device without & with feedback (Experimental): Participants will receive a Spire device with user-feedback switched off within 4 days of enrollment in the study (shipped within 2 business days after they finish enrollment survey). Participants will be given 4 days, after enrollment, to set up their device before the 2 weeks of baseline. The 2 week baseline will start 4 days after enrollment. After two weeks of baseline with user-feedback off (and a 3 day transition period), participants will turn on the user-feedback for the Spire device which would provide a relaxation aid for the participant for the 6 remaining weeks.
  Interventions: Device: Spire
- Muse device & spire device no feedback (Experimental): Participants in this group will also receive Spire device to assess two weeks of baseline stress levels (with user-feedback off). Participants will be given 4 days, after enrollment, to set up their device before the 2 weeks of baseline. The 2 week baseline will start 4 days after enrollment. After these two weeks, participants will continue to use the Spire device with user feedback off for the remaining 6 weeks while they use the Muse device to manage stress through meditation. They will receive the Muse device 3 days before the end of baseline period with set up instructions and will utilize the three last days of baseline to set up their Muse device, Meditation will begin at the end of baseline (week three) and will continue for the remaining 6 weeks.
  Interventions: Device: Spire; Device: Muse headband

INTERVENTIONS:
Device: Spire
Device: Muse headband
  Other Names: InteraXon
  Arms: Muse device & spire device no feedback

SUMMARY:
The goal of this study is to evaluate the effectiveness of Spire and Muse on stress management. The study will be implemented as a 2-arm randomized controlled pilot study to assess the effect of either device on stress management from the end of baseline to closeout.

DETAILED DESCRIPTION:
Both Muse and Spire are recent technologies that could improve our understanding of stress management and enhance quality of healthcare. The goal of this study is to evaluate if Spire and Muse help individuals self-manage stress. Spire has been designed as a discrete clip-on tracker that monitors changes in respiration rate. With the companion app, this device displays breathing rates in real time and alerts the user through push notification in times of tension. Studies show that controlled breathing reduces stress. On the other hand, Muse is a headset device that uses EEG (electroencephalogram) sensors that measures electric brain frequencies. Muse guides the user in a form of simplified meditation by giving feedback in real time (i.e. calm, neutral, active) and audio clues to improve concentration. Previous studies have shown that engaging in meditation has the potential to reduce anxiety and stress.

ELIGIBILITY:
Inclusion Criteria:

* Registered for Partners HealthCare Connected Health Symposium 2016
* Over 18 years old
* Able to read and speak English
* Own a smartphone and have internet connection
* Willing to wear a Spire device during all hours (except sleep)
* Willing to use the Muse device (Group 2 ONLY)
* Willing to participate in a research study and sign the consent form

Exclusion Criteria:

* Not Registered for Partners HealthCare Connected Health Symposium 2016
* Under 18 years old
* Not able to read and speak English
* Do not own a smartphone and have internet connection
* Not willing to wear a Spire device during all hours (except sleep)
* Not willing to use the Muse device (Group 2 ONLY)
* Not willing to sign the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen S, Janicki-Deverts D, Miller GE. Psychological stress and disease. JAMA. 2007 Oct 10;298(14):1685-7. doi: 10.1001/jama.298.14.1685. No abstract available. PMID 17925521
- [Background] Ellis JG, Gehrman P, Espie CA, Riemann D, Perlis ML. Acute insomnia: current conceptualizations and future directions. Sleep Med Rev. 2012 Feb;16(1):5-14. doi: 10.1016/j.smrv.2011.02.002. Epub 2011 May 18. PMID 21596596
- [Background] Kassel JD, Stroud LR, Paronis CA. Smoking, stress, and negative affect: correlation, causation, and context across stages of smoking. Psychol Bull. 2003 Mar;129(2):270-304. doi: 10.1037/0033-2909.129.2.270. PMID 12696841
- [Background] Herman JP. Neural pathways of stress integration: relevance to alcohol abuse. Alcohol Res. 2012;34(4):441-7. PMID 23584110
- [Background] Tully PJ, Baker RA, Turnbull D, Winefield H. The role of depression and anxiety symptoms in hospital readmissions after cardiac surgery. J Behav Med. 2008 Aug;31(4):281-90. doi: 10.1007/s10865-008-9153-8. Epub 2008 Apr 9. PMID 18398676
- [Background] Michels N, Sioen I, Braet C, Eiben G, Hebestreit A, Huybrechts I, Vanaelst B, Vyncke K, De Henauw S. Stress, emotional eating behaviour and dietary patterns in children. Appetite. 2012 Dec;59(3):762-9. doi: 10.1016/j.appet.2012.08.010. Epub 2012 Aug 20. PMID 22918173
- [Background] Edmondson D, Green P, Ye S, Halazun HJ, Davidson KW. Psychological stress and 30-day all-cause hospital readmission in acute coronary syndrome patients: an observational cohort study. PLoS One. 2014 Mar 12;9(3):e91477. doi: 10.1371/journal.pone.0091477. eCollection 2014. PMID 24621575
- [Background] Nerurkar A, Bitton A, Davis RB, Phillips RS, Yeh G. When physicians counsel about stress: results of a national study. JAMA Intern Med. 2013 Jan 14;173(1):76-7. doi: 10.1001/2013.jamainternmed.480. No abstract available. PMID 23403892
- [Background] Avey H, Matheny KB, Robbins A, Jacobson TA. Health care providers' training, perceptions, and practices regarding stress and health outcomes. J Natl Med Assoc. 2003 Sep;95(9):833, 836-45. PMID 14527051
- [Background] Paulus MP. The breathing conundrum-interoceptive sensitivity and anxiety. Depress Anxiety. 2013 Apr;30(4):315-20. doi: 10.1002/da.22076. Epub 2013 Mar 6. PMID 23468141
- [Background] Vlemincx E, Van Diest I, Van den Bergh O. A sigh following sustained attention and mental stress: effects on respiratory variability. Physiol Behav. 2012 Aug 20;107(1):1-6. doi: 10.1016/j.physbeh.2012.05.013. Epub 2012 May 23. PMID 22634279
- [Background] Grossman P, Niemann L, Schmidt S, Walach H. Mindfulness-based stress reduction and health benefits. A meta-analysis. J Psychosom Res. 2004 Jul;57(1):35-43. doi: 10.1016/S0022-3999(03)00573-7. PMID 15256293
- [Background] Carmody J, Baer RA. Relationships between mindfulness practice and levels of mindfulness, medical and psychological symptoms and well-being in a mindfulness-based stress reduction program. J Behav Med. 2008 Feb;31(1):23-33. doi: 10.1007/s10865-007-9130-7. Epub 2007 Sep 25. PMID 17899351
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Leon KA, Hyre AD, Ompad D, Desalvo KB, Muntner P. Perceived stress among a workforce 6 months following hurricane Katrina. Soc Psychiatry Psychiatr Epidemiol. 2007 Dec;42(12):1005-11. doi: 10.1007/s00127-007-0260-6. Epub 2007 Oct 11. PMID 17932611
- [Background] Gandek B, Ware JE, Aaronson NK, Apolone G, Bjorner JB, Brazier JE, Bullinger M, Kaasa S, Leplege A, Prieto L, Sullivan M. Cross-validation of item selection and scoring for the SF-12 Health Survey in nine countries: results from the IQOLA Project. International Quality of Life Assessment. J Clin Epidemiol. 1998 Nov;51(11):1171-8. doi: 10.1016/s0895-4356(98)00109-7. PMID 9817135
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- See also: 12. Morajevi, N, "You can't force calm: designing and evaluating respiratory regulating interfaces for calming technology" — http://dl.acm.org/citation.cfm?id=2380326

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In reference to comment [2] we had 126 participants that were enrolled in the study but only 125 that started the study. One participant that signed the consent form did not pass the eligibility criteria and therefore was not randomized into a study group and did not start the study.
Groups:
- Spire Device Without & With Feedback: Participants will receive a Spire device with user-feedback switched off within 4 days of enrollment in the study (shipped within 2 business days after they finish enrollment survey). Participants will be given 4 days, after enrollment, to set up their device before the 2 weeks of baseline. The 2 week baseline will start 4 days after enrollment. After two weeks of baseline with user-feedback off (and a 3 day transition period), participants will turn on the user-feedback for the Spire device which would provide a relaxation aid for the participant for the 6 remaining weeks.
  Spire
- Muse Device & Spire Device no Feedback: Participants in this group will also receive Spire device to assess two weeks of baseline stress levels (with user-feedback off). Participants will be given 4 days, after enrollment, to set up their device before the 2 weeks of baseline. The 2 week baseline will start 4 days after enrollment. After these two weeks, participants will continue to use the Spire device with user feedback off for the remaining 6 weeks while they use the Muse device to manage stress through meditation. They will receive the Muse device 3 days before the end of baseline period with set up instructions and will utilize the three last days of baseline to set up their Muse device, Meditation will begin at the end of baseline (week three) and will continue for the remaining 6 weeks.
  Spire
  Muse headband
Period: Overall Study
Arm/Group | Spire Device Without & With Feedback | Muse Device & Spire Device no Feedback
Started | 63 | 62
Completed | 53 | 56
Not Completed | 10 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spire Device Without & With Feedback | Muse Device & Spire Device no Feedback | Total
Number analyzed (Participants) | 63 | 62 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.85 (11.72) | 37.46 (13.51) | 37.15 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 41 | 40 | 81
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 5 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 49 | 52 | 101
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 61 | 57 | 118
  Spain | 1 | 0 | 1
  Australia | 1 | 1 | 2
  Canada | 0 | 3 | 3
  United Kingdom | 0 | 1 | 1
Employment Status [Count of Participants; unit: Participants]
  Employed | 51 | 52 | 103
  Unemployed | 1 | 0 | 1
  Student | 7 | 7 | 14
  Retired | 0 | 1 | 1
  Unknown | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Difference in Perceived Stress and Stress Resilience From Enrollment to Closeout
Description: The change of perceived stress and stress resilience within and between Group 1 and 2 from enrollment to closeout.
  The change of perceived stress is measured by the Perceived Stress Scale-14 (a validated psychological instrument of 14 items), each each rated on a 5 point scale(0-4) for measuring the respondent's perception of stress in the past month.The PSS-14 ranges from 0 to a high score of 56, with a higher score indicating more stress (worse outcome).
  The change of stress resilience is measured by the Connor-Davidson Stress Resilience Scale (25 items). It evaluates different aspects of stress coping ability that seeks to understand how well respondents would be able to buffer adverse conditions and cope with stress, each rated on a 5 point scale (0-4). The CD-RISC ranges from 0 to 100, with a higher score representing better stress resilience (a better outcome).
Time Frame: total of 8 weeks (2 weeks of baseline + 6 weeks of intervention)
Population: Adults over 18 who responded to a online advertisement
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spire Device Without & With Feedback | Muse Device & Spire Device no Feedback
Number analyzed (Participants) | 63 | 62
units on a scale
  Perceived Stress Scale at Closeout: number analyzed (Participants) | 46 | 62
  Perceived Stress Scale at Closeout | 20.24 (7.89) | 19.15 (8.92)
  Perceived Stress Scale at Enrollment: number analyzed (Participants) | 46 | 47
  Perceived Stress Scale at Enrollment | 23.59 (8.83) | 22.49 (8.63)
  Stress Resilience at Enrollment: number analyzed (Participants) | 44 | 48
  Stress Resilience at Enrollment | 68.25 (14.57) | 70.00 (12.39)
  Stress Resilience at Closeout: number analyzed (Participants) | 44 | 48
  Stress Resilience at Closeout | 69.5 (14.6) | 73.44 (13.34)

ADVERSE EVENTS:
Groups:
- Group 1: Participants will receive a Spire device with user-feedback switched off within 4 days of enrollment in the study (shipped within 2 business days after they finish enrollment survey). Participants will be given 4 days, after enrollment, to set up their device before the 2 weeks of baseline. The 2 week baseline will start 4 days after enrollment. After two weeks of baseline with user-feedback off (and a 3 day transition period), participants will turn on the user-feedback for the Spire device which would provide a relaxation aid for the participant for the 6 remaining weeks.
  Spire
- Group 2: Participants in this group will also receive Spire device to assess two weeks of baseline stress levels (with user-feedback off). Participants will be given 4 days, after enrollment, to set up their device before the 2 weeks of baseline. The 2 week baseline will start 4 days after enrollment. After these two weeks, participants will continue to use the Spire device with user feedback off for the remaining 6 weeks while they use the Muse device to manage stress through meditation. They will receive the Muse device 3 days before the end of baseline period with set up instructions and will utilize the three last days of baseline to set up their Muse device, Meditation will begin at the end of baseline (week three) and will continue for the remaining 6 weeks.
  Spire
  Muse headband
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/62
Other Adverse Events (participants affected / at risk) | 1/63 | 0/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=63) | Group 2 (N=62)
Minor Adverse Event (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — One study participant developed a rash on skin on the location on which the spire device was worn (chest, waist, underarm).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No